CLINICAL TRIAL: NCT02267733
Title: Study of High-dose Influenza Vaccine Efficacy by Repeated Dosing IN Gammopathy Patients (SHIVERING Trial)
Brief Title: Study of High-dose Influenza Vaccine Efficacy by Repeated Dosing In Gammopathy Patients
Acronym: SHIVERING
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1406014244
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Influenza; Gammopathy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Disease (Experimental): Patients not requiring anti-tumor therapy
  Interventions: Drug: Fluzone
- Disease Requiring Anti-tumor therapy (Experimental): Patients that have disease requiring anti-tumor therapy at any time
  Interventions: Drug: Fluzone

INTERVENTIONS:
Drug: Fluzone — Fluzone High-Dose will be administered with a planned booster at 30 days post initial administration
  Other Names: Fluzone High Dose

SUMMARY:
A Pilot Study utilizing high dose trivalent influenza vaccine dose in a booster dosing schedule for patients with monoclonal gammopathies stratified by disease status

DETAILED DESCRIPTION:
In this study, we will administer Fluzone® High-Dose vaccine with a planned booster to patients with monoclonal gammopathies (stratified by requirement for therapy) irrespective of age. All patients will receive an initial vaccine followed by a booster vaccine 30 days (+/- 7 days) later and will then be followed for outcomes until the end of flu season.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document
* Age >= 18 years at the time of signing the informed consent form
* Diagnosis of any monoclonal gammopathy; Monoclonal Gammopathy of Undetermined Significance (MGUS), asymptomatic/ active multiple myeloma, asymptomatic / active Waldenstrom Macroglobulinemia (WM)

Exclusion Criteria:

* An serious egg allergy or prior serious adverse reaction to an influenza vaccine
* Use of any other influenza vaccine for the 2014 to 2015 flu season
* Women who are pregnant or plan to become pregnant in the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of Disease Control | up to 10 months
  Lack of disease progression requiring therapy as measured by International Myeloma Working Group criteria

SECONDARY OUTCOMES:
Influenza related morbidity rate | up to 10 months
  Measure the rate of influenza related morbidity at the end of the flu season
Serologic Protection Rate after initial vaccine | 30 days post vaccine
  Evaluate rates of serologic protection (defined as HAI titer > 40) following initial vaccine dose
Serologic Protection Rate after initial vaccine | 30 days post booster
  Evaluate rates of serologic protection (defined as HAI titer > 40) following booster vaccine dose
T cell response | 30 day post initial vaccine
  Measurement of CD4+/CD8+, NK cells and influenza-specific T cell
T cell response | 30 day post booster
  Measurement of CD4+/CD8+, NK cells and influenza-specific T cell

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Branagan, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States